CLINICAL TRIAL: NCT00848952
Title: Performance of Imaging for the Diagnosis of Small Hepatocellular Carcinoma (< 3 cm)on Cirrhosis
Acronym: CHIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Christophe Aubé, University Hospital Angers
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHRC 2008-01
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

INTERVENTIONS:
Other: 3 imaging techniques are done — all patients have : MRI, CTscanner, enhanced contrast ultrasound

SUMMARY:
The purpose of this study is to evaluate 3 imaging techniques and their associations : MRI, CTscanner and enhanced contrast ultrasound for the diagnosis of small (< 3 cm) hepatocellular carcinoma for patients with cirrhosis.

DETAILED DESCRIPTION:
With the improvement of cirrhosis complications coverage, hepatocellular carcinoma (HCC) tend to become the main cause of mortality for cirrhotic patients. Currently, the incidence of the HCC increase in occidental country and hid global prognostic remain very bad. The main indication factor for a curative treatment is the size lesion.

Cirrhosis is the main risk factor for HCC occurence. In France, HCC screening has been establish for cirrhotic patients with hepatic ultrasound and alfa-fetoprotein measurement with the aim of detected HCC when the size allows a curative treatment.

When a nodule is discovered during the follow-up, HCC diagnosis is done following the recommendations of European Association for the Study of the Liver (AESL) in 2000, updated by the American Association for the Study of Liver Diseases (AASLD)in 2005. Diagnostic is function of nodule feature on one or two enhanced imaging techniques among CTscanner, MRI and enhanced contrast ultrasound.

This diagnostic strategy raises several questions. First, neither the most efficient dynamic imaging association for nodules from 1 to 2 cm, nor the most efficient imaging examination for nodules from 2 to 3 cm are known. Second, only few studies have been carried out about imaging semiology of the small hepatocellular carcinoma. Thus, the imprecisions of the present recommendations regarding the choice of the best examination technique and the difficulties in the diagnosis of benign or malignant nature for small nodule can lead to a bad management of these patients.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 hears
* presence of one or several nodules < 3 cm
* known or suspected cirrhosis

Exclusion Criteria:

* psychiatric disease
* contraindication to one of the 3 imaging examinations (CTscanner, MRI, enhanced contrast ultrasound
* patient already treated by chemoembolization
* recurrence on the coagulation zone of a nodule already treated by per-cutaneous tumour destruction
* presence of a tumour (> 3 cm) associated to the nodule
* pregnant woman or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Report of proportion of the positives truths and the positive wrong for an examination | one year

CONTACTS AND LOCATIONS:
Locations (19):
- France (19):
  - CHU Angers, Angers
  - Hôpital Saint-André, Bordeaux
  - Chu, Caen
  - hôpital Beaujon, Clichy
  - hôpital Henri Mondor, Créteil
  - Hôpital Du Bocage, Dijon
  - CHU, Grenoble
  - Hôpital de la croix rousse, Lyon
  - Hôpital E. Herriot, Lyon
  - Hôpital Saint Éloi, Montpellier
  - Hôpital Brabois, Nancy
  - Hôpital Hôtel Dieu, Nantes
  - hôpital archet II, Nice
  - Hôpital Saint Antoine, Paris
  - Hôpital Haut-Lévèque, Pessac
  - Hôpital Pontchaillou, Rennes
  - Hôpital Nord, Saint-Etienne
  - Hôpital Paul Brousse, Villejuif
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Paisant A, Vilgrain V, Riou J, Oberti F, Sutter O, Laurent V, Rodes A, Guiu B, Cassinotto C, Trillaud H, Bricault I, Michalak S, Bruno O, Ronot M, Aube C. Comparison of extracellular and hepatobiliary MR contrast agents for the diagnosis of small HCCs. J Hepatol. 2020 May;72(5):937-945. doi: 10.1016/j.jhep.2019.12.011. Epub 2019 Dec 21. PMID 31870951
- [Derived] Aube C, Oberti F, Lonjon J, Pageaux G, Seror O, N'Kontchou G, Rode A, Radenne S, Cassinotto C, Vergniol J, Bricault I, Leroy V, Ronot M, Castera L, Michalak S, Esvan M, Vilgrain V; CHIC Group. EASL and AASLD recommendations for the diagnosis of HCC to the test of daily practice. Liver Int. 2017 Oct;37(10):1515-1525. doi: 10.1111/liv.13429. Epub 2017 Apr 26. PMID 28346737